CLINICAL TRIAL: NCT02560883
Title: Clinical Research in Hairy Cell Leukemia: Surveillance and Documentation of Clinical Outcomes in a Rare Form of Adult Leukemia
Brief Title: Hairy Cell Leukemia Patient Data Registry
Acronym: HCL-PDR
Status: Recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Hairy Cell Leukemia Foundation (Other)
Responsible Party: Principal Investigator, Michael Grever, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-12194
Record Dates: First submitted 2015-08-20; First posted 2015-09-25 (Estimated); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Leukemia, Other
Keywords: Hairy Cell
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall objective is to develop a clinical data registry that can be used to facilitate research with the ultimate goal of reducing the morbidity and/or mortality and improving the quality of life of patients diagnosed or living with hairy cell leukemia. With approximately 1,000 new cases of this rare disease identified in the US each year, HCL represents 2% of all cases of leukemia in adults. Considering the rarity of this chronic leukemia, the Hairy Cell Leukemia Foundation (HCLF), in partnership with investigators from its Centers of Excellence, seeks to develop a registry to help researchers identify new trends in outcomes, recognize the most effective treatments, discover previously unknown complications of the disease, and design clinical trials for new therapies.

DETAILED DESCRIPTION:
This clinical registry is being established to collect de-identified information on this rare disease. The registry created by assimilation of de- identified coded patient data will centralize information that can be used to improve the management of the many complications of this disease and its treatment. This study is focused on collection of clinically and biologically meaningful endpoints across multiple institutions; as such, it is not focused on a specific set of hypotheses but will collect data that will facilitate such analyses. The investigators will collect information related to the symptoms and the clinical course of the disease, to the complications from the disease and its treatment, presence of minimal residual disease, frequency of relapse and subsequent management, data on novel molecular markers associated with the prognosis.

In conjunction with the Department of Bioinformatics at The Ohio State University, the investigators have created a system for safeguarding the confidentiality and the identity of all patients who agree to participate in this research registry. Each participating institution will be responsible for de-identification of the data, using software developed by The Ohio State University, Department of Biomedical Informatics, before it is used in the registry. Each institution will confidentially maintain a code for linking this information to an individual patient.

Each participating institution will have direct control over the data contained in the registry that is associated with their respective patient population. As a result of these measures, should a patient wish to withdraw from the registry, the responsible institution will be able to immediately remove all records related to that patient from the registry.

ELIGIBILITY:
Inclusion:

* Patients with classic hairy cell leukemia
* Patients with the variant of hairy cell leukemia.

Exclusion:

* Children are excluded from the study, since Hairy Cell Leukemia wasn't described in children.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be a multi-institutional, international project that will collate clinical information from patients with Hairy Cell Leukemia from participating institutions in the Hairy Cell Leukemia Foundation. Patients within the United States with HCL, who live in remote areas, without access to a HCLFCenter of Excellence, may voluntarily submit their name and contact information, through the Hairy Cell Leukemia Foundation website.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-01-02 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Surveillance | up to 25 years
  Establish a database of Hairy Cell Leukemia patients diagnosed or living in US to track Hairy Cell Leukemia disease course, patient reported outcomes, morbidity, and patient survival.

SECONDARY OUTCOMES:
Research | up to 25 years
  facilitate research with the ultimate goal of reducing the morbidity and/or mortality and improving the quality of life of patients diagnosed or living with hairy cell leukemia. Assess the number and type of infections recorded in patients following diagnosis and before therapy versus the infectious complications following administration of therapy for the disease. Identify and characterize patients at each participating institution with autoimmune complications associated with their diagnosis (e.g., polyarticular arthritis; immune cytopenias; vasculitis), and describe the response to immunosuppressive therapy. Collect data regarding treatment for hairy cell leukemia and its impact on the autoimmune complications of the disease.

OTHER OUTCOMES:
Contact | up to 25 years
  Offer two-way communication with patients by providing information regarding Hairy Cell Leukemia, opportunities to participate in tissue banking, observational, and therapeutic clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Grever, MD, Principal Investigator — The Ohio State University Comprehensive Cancer Center
Locations (6):
- United States (4):
  - University of Miami/Soffer Clinical Research Center, Miami, Florida
  - Mayo Clinic, Rochester, Minnesota
  - University of Rochester /Wilmot Cancer Institute, Rochester, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
- Peter MacCallum Cancer Center, Melbourne, Victoria, Australia
- Cancer Care Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- See also: Hairy Cell Leukemia Foundation — http://www.hairycellleukemia.org/